CLINICAL TRIAL: NCT00240370
Title: A Phase 3, Randomized, Double-Blind, Active-Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of BMS-298585 in Combination With Metformin Compared to Pioglitazone in Combination With Metformin in Type 2 Diabetics With Inadequate Glycemic Control on Metformin Alone
Brief Title: A Study to Evaluate Combining Metformin With Muraglitazar or Pioglitazone in Type 2 Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV168-025
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2008-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — muraglitazar

INTERVENTIONS:
Drug: Muraglitazar

SUMMARY:
The purpose of this study is to evaluate if type 2 diabetics who have inadequate glycemic control on metformin alone, have a similar, or not inferior, glycemic response when treated with the combination of muraglitazar and metformin compared to pioglitazone and metformin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetics
* HbA1c ≥7.0% and ≤10.0%,currently receiving a stable dose of metformin 1500 to 2550 mg/day for at least 6 weeks prior to screening were enrolled in this study.
* Fasting C-peptide ≥1.0 ng/mL
* BMI≤41 kg/m2 mean fasting serum trig. ≤600 g/dL

Exclusion Criteria:

* symptomatic type 2 diabetics with > 10% weight loss 3 months prior to study
* history of diabetic ketoacidosis, hyperosmolar nonketotic coma, insulin therapy, inability to take muraglitazar, pioglitazone, or metformin according to investigator brochure or labeling
* History of MI (myocardial infarction), coronary angioplasty or bypass graft(s), valvular disease or repair, unstable angina pectoris, transient ischemic attack (TIA), cerebrovascular attack, or cerebrovascular accident (CVA) within 6 months, congestive heart failure (NYHA Class III and IV, uncontrolled hypertension, history of, or renal disease, peripheral vascular disease (PVD), pulmonary disease, gastrointestinal disease, active liver disease or endocrine disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1159
Dates: Start 2003-10; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Compare change from basline in HbA1c after 24 weeks and 50 weeks of treatment with muraglitazar + metformin vs. pioglitazone + metformin

SECONDARY OUTCOMES:
Change in FPG from basline to W24, proportion of subjects receiving therapeutic response at W24, percent change of fasting lipid levels from baseline to W11/12, change in
hs-CRP from baseline to W24

CONTACTS AND LOCATIONS:
Locations (85):
- United States (70):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Columbiana, Alabama
  - Local Institution, Mesa, Arizona
  - Local Institution, Peoria, Arizona
  - Local Institution, Carlisle, Arkansas
  - Local Institution, Jonesboro, Arkansas
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Pine Bluff, Arkansas
  - Local Institution, Sherwood, Arkansas
  - Local Institution, Anaheim, California
  - Local Institution, Artesia, California
  - Local Institution, Encino, California
  - Local Institution, Encintas, California
  - Local Institution, Fresno, California
  - Local Institution, Long Beach, California
  - Local Institution, Los Angeles, California
  - Local Institution, Northridge, California
  - Local Institution, Denver, Colorado
  - Local Institution, Hamden, Connecticut
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Hollywood, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Miami, Florida
  - Local Institution, New Port Richie, Florida
  - Local Institution, Saint Cloud, Florida
  - Local Institution, West Palm Beach, Florida
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Evansville, Indiana
  - Local Institution, Lafayette, Indiana
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Shreveport, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Detroit, Michigan
  - Local Institution, Gulfport, Mississippi
  - Local Institution, St Louis, Missouri
  - Local Institution, Omaha, Nebraska
  - Local Institution, Endwell, New York
  - Local Institution, Cary, North Carolina
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Raleigh, North Carolina
  - Local Institution, Rudd, North Carolina
  - Local Institution, Statesville, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Bellbrook, Ohio
  - Local Institution, Maumee, Ohio
  - Local Institution, Thornville, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Portland, Oregon
  - Local Institution, Camp Hill, Pennsylvania
  - Local Institution, Melrose Park, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, West Chester, Pennsylvania
  - Local Institution, Youngwood, Pennsylvania
  - Local Institution, East Providence, Rhode Island
  - Local Institution, Charleston, South Carolina
  - Local Institution, Clinton, South Carolina
  - Local Institution, Memphis, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Carrollton, Texas
  - Local Institution, Corpus Christi, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Midland, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Lebanon, Virginia
  - Local Institution, Spokane, Washington
  - Local Institution, Tacoma, Washington
  - Local Institution, Bluefield, West Virginia
- Canada (7):
  - Local Institution, Red Deer, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Sarnia, Ontario
  - Local Institution, Bonaventure, Quebec
  - Local Institution, Drummondville, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Rimouski, Quebec
- Mexico (6):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Mexico, Durango
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Cuernavaca, Morelos
- Puerto Rico (2):
  - Local Institution, Aguas Buenas
  - Local Institution, Ponce